CLINICAL TRIAL: NCT02976051
Title: DAHANCA 33: Functional Image Guided Dose-escalated Radiotherapy to Patients With Hypoxic Squamous Cell Carcinoma of the Head and Neck
Brief Title: DAHANCA 33: Image Guided Dose-escalated Radiotherapy to Patients With Hypoxic HNSCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Head and Neck Cancer Group (Network)
Responsible Party: Principal Investigator, Jens Overgaard, Professor, MD DMSc, Danish Head and Neck Cancer Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAHANCA 33
Record Dates: First submitted 2016-11-22; First posted 2016-11-29 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Locally Advanced Head and Neck Cancer; Radiotherapy; Hypoxic Radioresistance
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with HART-CN (Experimental): HART-CN: Hyperfractionated accelerated radiotherapy with weekly concommitant cisplatin and nimorazole
  Interventions: Radiation: HART-CN

INTERVENTIONS:
Radiation: HART-CN — HART-CN: Hyperfractionated accelerated radiotherapy with weekly concommitant cis-platin and daily nimorazole

SUMMARY:
Aim: To improve curability of radiotherapy in HNSCC patients identified by hypoxic FAZA-PET scanning

DETAILED DESCRIPTION:
Prospective phase II study aiming to improve the outcome in hypoxic resistent patients identified by FAZA-PET.

Inclusion:

Patients must fulfill the following:

Positive hypoxic FAZA-PET Scanning (as described in DAHANCA 24 - see citation) Stage III-IV, Squamous cell carcinoma of the larynx, pharynx or oral cavity (HPVneg (oropharynx) Indication for hyperfractionated accelerated radiotherapy with concommitant cis-platin and nimorazole

ELIGIBILITY:
Inclusion Criteria:

* Stage III-IV larynx, pharynx, oral cavity
* Hypoxic FAZA-PET positive
* Indication for primary radio-chemotherapy
* Informed consent

Exclusion Criteria:

* HPV positive oropharynx cancer
* Primary surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Loco-regional failure | Year 3
  loco-regional failure defined as persistent or recurrent disease in tumor and/or regional lymphnode sites (within the radiotherapy treated volume). The primary endpoint did not include the effect of a successful procedure with salvage surgery (no primary neck dissection was allowed).

SECONDARY OUTCOMES:
Overall survival | Year 3
  Death from all causes
Acute radiation related morbidity | Month 3
Late radiation related morbidity | Year 3
Disease-specific death | Year 3
  Disease-specific death is defined as death from or with the cancer in question;

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Experimental Clinical Oncology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mortensen LS, Johansen J, Kallehauge J, Primdahl H, Busk M, Lassen P, Alsner J, Sorensen BS, Toustrup K, Jakobsen S, Petersen J, Petersen H, Theil J, Nordsmark M, Overgaard J. FAZA PET/CT hypoxia imaging in patients with squamous cell carcinoma of the head and neck treated with radiotherapy: results from the DAHANCA 24 trial. Radiother Oncol. 2012 Oct;105(1):14-20. doi: 10.1016/j.radonc.2012.09.015. Epub 2012 Oct 16. PMID 23083497